CLINICAL TRIAL: NCT07181096
Title: Study of Frailty Among Renal Transplant Recipients, Its Relation to Chronic Renal Allograft Dysfunction
Brief Title: Frailty Among Renal Transplant Recipients and Relation to Chronic Allograft Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Associate professor, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: frailty in renal transplant
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Frailty; Renal Transplant
Keywords: Frailty; renal transplant recipient; chronic allograft dysfunction
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- renal transplant patients (Experimental): patients will be subjected to:
  1. Assessment of frailty by Clinical Frailty Scale.
  2. Assessment of nutritional status using Patient Generated Subjective Global Assessment (PG-SGA).
  3. Comorbidity assessment using Charlson comorbidity score.
  4. Six minutes walk test.
  5. Muscle strength assessment using hand grip strength (HGS) dynamometer.
  Interventions: Diagnostic Test: assessment of frailty

INTERVENTIONS:
Diagnostic Test: assessment of frailty — This study is a prospective cross-sectional study to assess the prevalence of frailty among 80 cases of renal transplanted patients.
  Specific tests will include:
  1. Assessment of frailty by Clinical Frailty Scale.
  2. Assessment of nutritional status using Patient Generated Subjective Global Assessment (PG-SGA).
  3. Comorbidity assessment using Charlson comorbidity score.
  4. Six minutes walk test.
  5. Muscle strength assessment using hand grip strength (HGS) dynamometer.

SUMMARY:
The aim of the study is to assess prevalence of frailty among renal transplant recipients in Alexandria University Hospitals and to study the relation between frailty and chronic allograft dysfunction.

DETAILED DESCRIPTION:
With respect to correlates of frailty, although higher comorbidity burden is also a risk factor for frailty among KT candidates, frailty can also occur in the setting of lower comorbidity burdens. Diabetes and serum albumin concentration are also associated with frailty among prevalent dialysis patients.

In addition, individuals with CKD and ESKD who are frail are also more likely to have cognitive impairment and sarcopenia, or low muscle mass, than their non-frail counterparts

ELIGIBILITY:
Inclusion Criteria:

* Renal transplanted patients with GFR more than 30

Exclusion Criteria:

* Mentally or physically unfit patients.
* Amputation of lower limb.
* Active neoplasia, chronic liver disease, previous immunological disease.
* Psychiatric disorders.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of frailty | 30 days
  by Clinical Frailty Scale.

SECONDARY OUTCOMES:
Assessment of nutritional status | 30 days
  using Patient Generated Subjective Global Assessment (PG-SGA)
Comorbidity assessment | 30 days
  using Charlson comorbidity score
Muscle strength assessment | 30 days
  using hand grip strength (HGS) dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed mamdouh Elsayed, MD, Principal Investigator — Associate professor; salah saed naga, MD, Principal Investigator — professor; hala seddik elwakil, MD, Study Chair — professor; dalia ezzat saleh, MBBCH, Study Chair — resident
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lorenz EC, Cosio FG, Bernard SL, Bogard SD, Bjerke BR, Geissler EN, Hanna SW, Kremers WK, Cheng Y, Stegall MD, Cheville AL, LeBrasseur NK. The Relationship Between Frailty and Decreased Physical Performance With Death on the Kidney Transplant Waiting List. Prog Transplant. 2019 Jun;29(2):108-114. doi: 10.1177/1526924819835803. Epub 2019 Mar 17. PMID 30879429
- [Background] Alfieri C, Malvica S, Cesari M, Vettoretti S, Benedetti M, Cicero E, Miglio R, Caldiroli L, Perna A, Cervesato A, Castellano G. Frailty in kidney transplantation: a review on its evaluation, variation and long-term impact. Clin Kidney J. 2022 May 24;15(11):2020-2026. doi: 10.1093/ckj/sfac149. eCollection 2022 Nov. PMID 36325001
- [Background] Quint EE, Zogaj D, Banning LBD, Benjamens S, Annema C, Bakker SJL, Nieuwenhuijs-Moeke GJ, Segev DL, McAdams-DeMarco MA, Pol RA. Frailty and Kidney Transplantation: A Systematic Review and Meta-analysis. Transplant Direct. 2021 May 18;7(6):e701. doi: 10.1097/TXD.0000000000001156. eCollection 2021 Jun. PMID 34036171